CLINICAL TRIAL: NCT04242160
Title: Prospective Randomized Trial of Standard Left Anterolateral Thoracotomy vs Modified Bilateral Clamshell Thoracotomy Performed by Emergency Physicians
Brief Title: Comparison of Two Resuscitative Thoracotomy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency); United States Air Force En Route Care Research Center (Unknown); Centre for Emergency Health Sciences (Unknown); Barts & The London NHS Trust (Other); The Institute of Pre-Hospital Care at London's Air Ambulance (Unknown); US Air Force 711th Human Performance Wing (Unknown)
Responsible Party: Principal Investigator, Derek J Brown, MD, Emergency Medicine Physician, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C.2017.172e
Record Dates: First submitted 2020-01-19; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Emergencies; Trauma; Procedural Training; Thoracotomy
MeSH Terms: conditions — Emergencies; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants were randomized to the order of intervention. After completing the first RT technique assigned, participants complete the alternative RT technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Clamshell Thoracotomy First (Experimental): Participants randomized to perform the MCT first, then cross over to the perform the alternate LAT.
  Interventions: Other: Modified Clamshell Thoracotomy; Other: Left Anterolateral Thoracotomy
- Left Anterolateral Thoracotomy First (Active Comparator): Participants randomized to perform the LAT first, then cross over to the perform the alternate MCT.
  Interventions: Other: Modified Clamshell Thoracotomy; Other: Left Anterolateral Thoracotomy

INTERVENTIONS:
Other: Modified Clamshell Thoracotomy — Participants received standardized training on performing a MCT and LAT. Participants then performed the procedures on a fresh human cadaver model.
Other: Left Anterolateral Thoracotomy — Participants received standardized training on performing a MCT and LAT. Participants then performed the procedures on a fresh human cadaver model.

SUMMARY:
Resuscitative thoracotomy (RT) is a life saving procedure for patients who have suffered cardiac arrest or are at significant risk of cardiac arrest following significant trauma. The procedure is ideally performed by a surgeon, but in some circumstance must be performed by non-surgical specialists such as Emergency Medicine physicians. The purpose of this study was to evaluate the optimal RT technique taught to non-surgical specialists in an educational human cadaver lab. The objective was to compare time to successful completion of two different RT techniques; (1) Left Anterolateral Thoracotomy (LAT) and (2) Modified Clamshell Thoracotomy (MCT). The investigators hypothesized that the non-surgical specialist time to successful completion for the MCT would be shorter than for the LAT.

DETAILED DESCRIPTION:
The investigators conducted a randomized crossover trial of two resuscitative thoracotomy techniques performed by Emergency Medicine (EM) physicians using a fresh human cadaver model. The purpose was to identify the ideal technique to be taught to non-surgical specialists in a training lab setting. The two techniques compared were the Left Anterolateral Thoracotomy (LAT), commonly taught to EM physicians in the United States, and the Modified Clamshell Thoracotomy (MCT) taught by London's Air Ambulance. The investigators hypothesized that the non-surgical specialists time to successful completion of the RT would be faster when performing the MCT compared to the LAT.

The investigators conducted this study at a large level 1 trauma center with an Emergency Medicine residency program and recruited Emergency Medicine residents and staff physicians to participate. Participants were trained on the MCT as performed by LAA and reviewed the LAT technique in a standardized fashion. Participants were then randomized to order of intervention, and conducted each procedure on a separate fresh human cadaver. Participants were evaluated on time to successful completion of the procedure, successful completion of procedural steps, and identification of anatomy. Cadaver specimens were examined for iatrogenic injuries. Participants then completed a standardized survey regarding each procedure.

ELIGIBILITY:
Inclusion Criteria:

* licensed physician
* emergency medicine residency trainee or graduate
* privileged provider at SAMMC

Exclusion Criteria:

- unwilling to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Time to successful completion of RT procedure | During procedure on data collection date
  Time participant took to complete a successful RT procedure. Success includes (1) successful delivery of the heart and (2) successful cross-clamp of the descending thoracic aorta. Success determined by general surgeon observer. Time start from command "go" until participant verbalizes delivery of the heart and cross-clamp of the aorta.

SECONDARY OUTCOMES:
Successful delivery of the heart defined as exposure and inspection of all surfaces | During procedure on data collection date
  Determined by General Surgeon observer
Successful descending thoracic aorta cross-clamp defined as 100% occlusion of the descending aorta with a vascular clamp | During procedure on data collection date
  Determined by General Surgeon observer
Time to delivery of the heart defined as exposure and inspection of all surfaces | During procedure on data collection date
  time from command "go" to subject verbalizing delivery of heart
Time to descending thoracic aorta cross clamp defined as 100% occlusion of the descending aorta with a vascular clamp | During procedure on data collection date
  total elapsed time from command "go" to subject verbalizing successful cross-clamping of the descending thoracic aorta
Occurrence of iatrogenic injuries | During procedure on data collection date
  Injury to phrenic nerve, esophagus, lung, heart or other anatomical structure as identified by a General Surgeon AI.
Successful identification of anatomy | During procedure on data collection date
  Successful identification of the phrenic nerve, right atrium, left atrium, right ventricle, left ventricle, pulmonary hilum, descending thoracic aorta, and esophagus.
Subject Questionnaire | During procedure on data collection date
  Procedural ease, comfort, view, equipment comfort and preference.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newberry R, Brown D, Mitchell T, Maddry JK, Arana AA, Achay J, Rahm S, Long B, Becker T, Grier G, Davies G. Prospective Randomized Trial of Standard Left Anterolateral Thoracotomy Versus Modified Bilateral Clamshell Thoracotomy Performed by Emergency Physicians. Ann Emerg Med. 2021 Mar;77(3):317-326. doi: 10.1016/j.annemergmed.2020.05.042. Epub 2020 Aug 15. PMID 32807537